CLINICAL TRIAL: NCT06182800
Title: A Prospective Study of Adebrelimab Combined With Bevacizumab and Docetaxel in the Treatment of Advanced Non-Squamous Non-small Cell Lung Cancer After Progression on First-line Immunotherapy
Brief Title: Adebrelimab Combined With Bevacizumab and Docetaxel for Advanced Non-Squamous Non-small Cell Lung Cancer After Progression on First-line Immunotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Principal Investigator, Yinghua Ji, chief of oncology, The First Affiliated Hospital of Xinxiang Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY202319
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab Combined with Bevacizumab and Docetaxel (Experimental): Adebrelimab: 1200 mg Adebrelimab is given on day 1 of each cycle, with 1 dosing cycle every 3 weeks. The dosing time window may be ±5 days, but within 72 hours before each dose, subjects must complete an examination including all clinically necessary tests to assess tolerability of continued dosing, in addition to imaging. Subjects are also advised to remain in the hospital for observation 72 hours after the first dose.
  Bevacizumab: 7.5 mg/kg Bevacizumab administered intravenously on day 1 of each cycle, with 1 dosing cycle every 3 weeks.
  Docetaxel: 60-75 mg/m2 Docetaxel is given on days 1 of each cycle by intravenous infusion for 1 dosing cycle every 3 weeks.
  Interventions: Drug: Adebrelimab Combined with Bevacizumab and Docetaxel

INTERVENTIONS:
Drug: Adebrelimab Combined with Bevacizumab and Docetaxel — Adebrelimab: 1200 mg Adebrelimab is given on day 1 of each cycle, with 1 dosing cycle every 3 weeks. The dosing time window may be ±5 days, but within 72 hours before each dose, subjects must complete an examination including all clinically necessary tests to assess tolerability of continued dosing, in addition to imaging. Subjects are also advised to remain in the hospital for observation 72 hours after the first dose.
  Bevacizumab: 7.5 mg/kg Bevacizumab administered intravenously on day 1 of each cycle, with 1 dosing cycle every 3 weeks.
  Docetaxel: 60-75 mg/m2 Docetaxel is given on days 1 of each cycle by intravenous infusion for 1 dosing cycle every 3 weeks.

SUMMARY:
This study is a prospective, single-arm, multicenter, phase II clinical study to observe and evaluate the efficacy and safety of adebrelimab in combination with bevacizumab and docetaxel in patients with advanced non-squamous NSCLC after progression on first-line immunotherapy.

DETAILED DESCRIPTION:
The study consisted of a screening period (no more than 4 weeks after patients signed informed consent until enrollment, with imaging assessments allowed to be archived within 4 weeks prior to enrollment), a treatment period (treatment termination defined as discontinuation of treatment for any reason, or withdrawal from the study for any reason), a safety follow-up period, and a survival follow-up period.

Screening period:

Patients were required to undergo a screening evaluation to determine their eligibility for the study within 4 weeks prior to enrollment.

Patients eligible for the study receive adebrelimab, 1200 mg, Intravenous infusion, every 3 weeks (Q3W) + bevacizumab, 7.5 mg/kg, Intravenous infusion, Q3W +docetaxel 60-75 mg/m2, D1, Intravenous infusion, Q3W. docetaxel for 4 cycles, adebrelimab, bevacizumab use to progressive disease (PD), intolerable toxicity, patient withdrawal of informed consent, investigator decision to discontinue study treatment.

Treatment period:

Patients eligible for study enrollment were given medication sequentially on day 1 of each cycle, with a dosing window of ±5 days, and patients were required to complete various examinations including vital signs, height and weight, physical examination, laboratory tests, and physical status scores to assess tolerance for continued treatment. The specific examinations and requirements for each visit are shown in the study flow chart.

End of treatment:

End of treatment is defined as confirmation of disease progression or withdrawal from the study and requires an end-of-treatment visit ±5 days from the time of the decision to discontinue treatment and/or withdraw from the study.

Safety follow-up. Safety follow-up visits will be conducted within 30±7, 60±7 days, and 90±7 days after the last dose.

Survival follow-up. Survival follow-up will be conducted every 3 months after safety follow-up and telephone follow-up is acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily enrolled in this study and signed the Informed Consent Form (ICF).
2. age ≥ 18 years and both sexes
3. patients with metastatic or recurrent stage IV non-squamous NSCLC (AJCC 8th edition Tumor Node Metastasis (TNM) stage) proven by histopathological or cytopathological diagnosis, mainly including adenocarcinoma, large cell lung cancer, adenocarcinoma with squamous differentiation or adenosquamous carcinoma with predominantly adenocarcinoma component may also be enrolled if eligible by study assessment.
4. objective imaging progression (RECIST v1.1 assessment) after subjects have received a first-line regimen containing immune checkpoint inhibitor therapy.
5. the immune checkpoint inhibitor-containing therapy PFS of ≥ 6 months on first- line therapy.
6. imaging evaluation (CT or MRI) with at least one measurable target lesion (according to RECIST v1.1) within 4 weeks prior to enrollment.
7. an ECOG PS score of 0-1 within 4 weeks prior to enrollment.
8. an expected survival of ≥ 12 weeks.
9. Adequate function of vital organs
10. Non-surgical sterilization or female patients of childbearing age must have a negative serum pregnancy test within 7 days prior to the first dose and must be non-lactating. Female patients of childbearing age or male patients whose partners are women of childbearing age must agree to use highly effective methods of contraception during the study period and for 6 months after the last administration of the study drug.

Exclusion Criteria:

1. patients with other pathological tissue types of non-small cell lung cancer (including squamous cell carcinoma, mixed non-small cell and small cell lung cancer, and predominantly squamous adenosquamous carcinoma of the lung)
2. patients with known EGFR-sensitive mutations (19Exon del/21Exon L858R), positive ALK/ROS1 fusion.
3. patients with imaging showing signs of tumor invasion into the great vessels, where the tumor has completely approached, encircled, or invaded the lumen of a great vessel (e.g., pulmonary artery or superior vena cava)
4. patients with hypertension whose blood pressure is not satisfactorily controlled by antihypertensive medication (sitting systolic blood pressure > 150 mmHg, or diastolic blood pressure > 100 mmHg), previous hypertensive crisis or hypertensive encephalopathy.
5. those with a known hereditary bleeding tendency or coagulation disorders; those who have received full-dose anticoagulant or thrombolytic therapy within 10 days prior to enrollment, or those who have taken non-steroidal anti-inflammatory drugs with platelet inhibitory effects within 10 days prior to enrollment (except for prophylactic use of low-dose aspirin (≤325 mg/day)).
6. had a hemoptysis of 2nd degree or greater with a single hemoptysis of ≥1/2 teaspoon (2.5 ml) within 3 months prior to enrollment thrombosis in the 6 months
7. prior to enrollment and an arterial/venous thrombotic event within 1 year prior to screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism.
8. those with severe vascular lesions (including aneurysms or arterial thrombosis requiring surgical treatment) within 6 months prior to enrollment
9. late first-line treatment with anti-angiogenic agents, including but not limited to bevacizumab, apatinib, anlotinib, ramucirumab, lenvatinib, etc.; treatment with docetaxel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-12-27 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | 6 months
  6-Month PFS Rates for Adebrelimab Combined with Bevacizumab and Docetaxel in Patients with Advanced Non-Squamous NSCLC Progressed by First-Line Immunotherapy Evaluated by Investigators

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
  PFS is defined as the time elapsed between the start of treatment and the first sign of disease progression or death from any cause.
Over survival (OS) | up to 18 months
  OS is defined as the time elapsed between the initiation of treatment and mortality from any cause.
objective response rate (ORR) | up to 12 months
  Number of cases with completed/partial response after treatment as a percentage of evaluable cases.

IPD SHARING:
Plan to Share IPD: No